CLINICAL TRIAL: NCT05756023
Title: IVF\ICSI Outcome in Women With Polycystic Ovary Syndrome Compared With Non Polycystic Ovary Syndrome Women
Brief Title: IVF\ICSI Outcome in Women With Polycystic Ovary Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Islam Mahfouz
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCOs Patients (Active Comparator): To compare the pregnancy rate at IVF / ICSI cycles in patients with PCOs
  Interventions: Procedure: the pregnancy rate at IVF / ICSI cycles
- Non PCOs Patients (Active Comparator): To compare the pregnancy rate at IVF / ICSI cycles in patients with without PCOs
  Interventions: Procedure: the pregnancy rate at IVF / ICSI cycles

INTERVENTIONS:
Procedure: the pregnancy rate at IVF / ICSI cycles — To study and compare other parameters between the PCOS and non PCOS group, and inside the PCOS group itself eg ; patients with PCOS who have ovarian drilling and non drilling PCOS

SUMMARY:
Polycystic ovarian syndrome (PCOS) occurs in 5% to 10% of all women of reproductive age and 50% of women who present with sub-fertility due to anovulatory infertility . Clear diagnostic criteria for this condition were identified at the consensus meeting of the European Society of Human Reproduction and Embryology and the American Society for Reproductive Medicine .

DETAILED DESCRIPTION:
Sub-fertile women with PCOS will usually benefit from conventional treatments, such as lifestyle changes, ovulation induction, or laparoscopic ovarian drilling, but some will ultimately need assisted reproductive techniques, either if they will need or if they wish, such as controlled ovarian hyperstimulation and IVF.

In these cases, controlled ovarian hyperstimulation is closely related to high drug costs, need for daily injections and frequent monitoring, whereas it sometimes results in an increased rate of cycle cancellations and potential life threatening complications due to ovarian hyperstimulation syndrome and in the retrieval of immature oocytes, leading to poor fertilization and lower cleavage, pregnancy, and live birth rates compared to the conventional IVF cycles ,although this has not been confirmed by other studies .

In addition, ovulation induction is associated with a high risk of multiple pregnancies due to multiple follicular development, so that it has to be individualized and closely monitored.

In-vitro fertilization (IVF) is a common therapeutic modality used in infertile women. IVF has different success rates in different subgroups of patients.

It is necessary to alter the common standard protocols to overcome the potential obstacles in some populations of patients and achieve the best results . Obesity with PCOS status of patient may decrease the fertilization rate and clinical pregnancy chance after IVF (probably by decreasing the oocyte count and increasing the gonadotropin resistance); however, the results of different studies are conflicting

ELIGIBILITY:
Inclusion Criteria:

* Oligo-ovulation or anovulation.
* Clinical and/or biochemical hyper androgenesim.
* Polycystic ovaries.

Exclusion Criteria:

1. Androgen-secreting tumors (ovarian or adrenal).
2. Adult-onset congenital adrenal hyperplasia.
3. Thyroid diseases.
4. Cushing's syndrome.
5. Diabetes Mellitus.
6. recurrent ICSI failure
7. endocrine, hematologic and autoimmune disorders
8. Non chromosomal and genetic abnormalities
9. Major uterine anomalies, bad surgical history, sever endometriosis, , hydrosalpinx, uterine fibroids
10. Azospermia

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | From baseline to 15 days after the embryo transfere day.
  To compare the pregnancy rate at IVF / ICSI cycles between women with PCOS and non PCOS women

CONTACTS AND LOCATIONS:
Overall Officials: Momen Kamel, Professor, Study Chair — Assiut University, Faculty of medicine, Assuit.
Locations (1):
- Assuit University hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No